CLINICAL TRIAL: NCT01833559
Title: Impact of Blood Glucose at the First Trimester of Pregnant Women With Gestational Diabetes on Maternal and Fetal Outcomes and Metabolic Disorders: a Multi-central Prospective Cohort Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zilian Wang, Doctor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GDMTEST-5010-00; GDMTEST-5010-01 (Registry Identifier: Gynecology and obstetrics department of the 1st affiliated hospital of Sun Yat-sen University); GDMTEST-5010-02 (Registry Identifier: Gynecology and obstetrics department of the 3rd affiliated hospital of Sun Yat-sen University); GDMTEST-5010-03 (Registry Identifier: Guangdong women and children hospital); GDMTEST-5010-04 (Registry Identifier: Guangzhou women and children hospital)
Record Dates: First submitted 2013-04-10; First posted 2013-04-17 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Insulin; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Incidence of GDM (Other): Dietary control will be suggested to patients if their fasting blood glucose is between 5.1 mmol/L and 7.0 mmol/L. If feast blood glucose is over 7.0 mmol/L, the patient will be hospitalized.
  Interventions: Dietary Supplement: Dietary control; Drug: Insulin
- Gestational outcomes (Other): Dietary control will be suggested to patients if their fasting blood glucose is between 5.1 mmol/L and 7.0 mmol/L. If feast blood glucose is over 7.0 mmol/L, the patient will be hospitalized.
  Interventions: Dietary Supplement: Dietary control; Drug: Insulin
- Metabolic disorder (Other): Dietary control will be suggested to patients if their fasting blood glucose is between 5.1 mmol/L and 7.0 mmol/L. If feast blood glucose is over 7.0 mmol/L, the patient will be hospitalized.
  Interventions: Dietary Supplement: Dietary control; Drug: Insulin

INTERVENTIONS:
Dietary Supplement: Dietary control
Drug: Insulin — If feast blood glucose is over 7.0 mmol/L, the patient will be hospitalized and insulin will be used. The kind of insulin used depends on the need of patients.
  Other Names: Novolin R; Novolin N; Novolin 30R; Novolin 50R

SUMMARY:
The study is to investigate the impact of blood glucose management at the first trimester of pregnant women with gestational diabetes on the maternal and fetal outcomes and metabolic disorder.

DETAILED DESCRIPTION:
Gestational diabetes(GDM) is the glucose metabolic disorder that first diagnosed during pregnancy. With the development of social economy and the improvement of life, the incidence of GDM increases to a level of 18-20% year by year. High blood glucose has a strong relationship with many adverse maternal and fetal outcomes, but also influences their metabolism including the increase of susceptibility of maternal type 2 diabetes and risk of fetal type 2 diabetes, obesity, coronary heart disease, etc. And therefore, it is significant to screening and managing maternal blood glucose to prevent maternal and fetal adverse outcomes and metabolic disorder.

This multi-central prospective cohort study is supposed to study the pregnant women whose fasting blood glucose is slightly increased (between 5.1 mmol/L and 7.0 mmol/L) at the first gestational trimester. The aim of this study is to answer the scientific questions bellow: whether interventions to whom the blood glucose is slightly increased can

1. decrease the incidence of GDM at the second gestational trimester;
2. improve gestational outcomes;
3. decrease the incidence of temporal and distant metabolic disorder of mother and her child.

The result will provide scientific evidence for improving the gestational outcomes of GDM women and preventing metabolic disorder of their child during adolescence and adult period.

ELIGIBILITY:
Inclusion Criteria:

* regular antenatal examination from the first trimester;
* accurate left mentoposterior(LMP) verified by ultrasonography(USG);
* fasting blood glucose level between 5.1 mmol/L and 7.0 mmol/L.

Exclusion Criteria:

* younger than 18 years old;
* do not give birth in the research centers above;
* LMP is undefined and lack of USG during 6-14 gestational weeks;
* multiple pregnancy;
* non-natural pregnancy(including intrauterine insemination(IUI), in-vitro fertilization and embryo transfer(IVF-ET), etc);
* diagnosed DM before pregnancy;
* with hepatitis B virus, hepatitis C virus, HIV infection;
* taking drugs including glucocorticoid, diuretic, angiotensin-converting enzyme inhibitor/angiotensin II receptor blocker(ACEI/ARB), etc.
* complicated with diseases that affect glucose metabolism such as hyperthyroidism and so on.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2012-06; Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of GDM at the second gestational trimester | at the second gestational trimester(about 24-28 gestational weeks)
  The results of oral glucose tolerance test(OGTT) at the second gestational trimester(about 24-28 gestational weeks) which is used to diagnose GDM will be recorded to analysis the incidence of GDM at the second gestational trimester.

SECONDARY OUTCOMES:
Gestational outcomes | After delivery
  The adverse gestational outcomes will be recorded. For example: GDM, preeclampsia,fetal growth restriction(FGR),and so on.

OTHER OUTCOMES:
The incidence of temporal and distant metabolic disorder of mother | 2 months to 1 year after delivery
  After about 2 months after delivery when mother comes back for postpartum follow-up, some tests will be done, such as regular blood test,blood glucose(fasting and 2 hours after meal), urine regular test and so on.
Child growth measures | 2 months to 1 year after delivery
  Children's body weight and height will be firstly recorded when their mothers come back for postpartum follow-ups at about 2 months after delivery by asking them or measure their children on the spot if they take their children with them.
  And the growth measures of children will be recorded for the second time by asking them via telephone at about 1 year after delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology and obstetrics department of the 1st affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China